CLINICAL TRIAL: NCT01803581
Title: A Randomized, Controlled, Investigator-blinded, Comparative Study to Evaluate the Safety and Efficacy of Product X92001327 vs RID Shampoo in Subjects With Head Lice
Brief Title: A Study to Evaluate the Safety and Efficacy of Product X92001327 vs RID Shampoo in Subjects With Head Lice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OYS004-0013
Record Dates: First submitted 2013-02-12; First posted 2013-03-04 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-11

CONDITIONS: Head Lice

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- X92001327 (Experimental): the X92001327 product is a lotion to be applied on dry hair for 15 minutes and then washed out using shampoo. The product is to be applied on Day 0 and repeated again on Day 7.
  Interventions: Other: X92001327
- RID shampoo (Active Comparator): The RID shampoo is to be applied on dry the hair for 10 minutes and then rinsed out with water. the product is to be applied on Day 0 and repeated again on Day 7.
  Interventions: Other: RID shampoo

INTERVENTIONS:
Other: X92001327
  Arms: X92001327
Other: RID shampoo
  Arms: RID shampoo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of an insecticide-free head lice product with that of a pyrethrum-based product.

DETAILED DESCRIPTION:
The primary objective of the study was to compare the safety and efficacy of X92001327 versus RID in subjects with head lice. The subjects received a single application on Day 0 of either X92001327 or RID shampoo based on the randomization schedule. A repeat application of the test product was administered on Day 7. Subjects visited the clinic four times: on Day 0, Day 1, Day 7 and Day 10.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 1 at the time of signing the informed consent or giving assent
* Have an active head lice infestation of at least 5 live lice and 5 viable nits
* subject must be capable of understanding and providing written informed consent
* agree not to use any other pediculicides or medicated hair grooming products for the duration of the study
* agree not to use a lice comb during the study
* the parent or guardian of a child must be willing to have other family members screened for head lice.
* have a single place of residence

Exclusion Criteria:

* used any form of head lice treatment whether prescription or over the counter or home remedy at least four weeks prior to their screening visit
* used any topical medication of any kind for a period of 48 hours prior to the screening visit
* individuals on systemic or topical drugs or medications, including systemic antibiotics, which in the opinion of the investigative personnel may interfere with the study results
* has a history of allergy or hypersensitivity to ragweed, hydrocarbons, sesame oil, perfume or any ingredient in either test product
* individuals with any visible skin/scalp condition at the treatment site which, in the opinion of the investigative personnel will interfere with the evaluation of the test product
* individuals who, in the opinion of the investigative personnel do not understand the subject requirements for study participation and/or may be likely to exhibit poor compliance with the required visits
* females who are pregnant or nursing
* patients that have taken trimethoprim or a combination of sulfamethoxazole at evaluation or during the previous 4 weeks
* subjects with hair longer than mid back

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03-05 (Actual); Primary Completion 2013-06-20 (Actual); Study Completion 2013-08-12 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects lice free at the end of the study (Day 10) | Day 10
  Primary objective of this study was the cure rate (%) in each treatment group, following two applications (day 0 and day 7) of the specific test product, as assessed on the last evaluation visit (day 10).

SECONDARY OUTCOMES:
The proportion of subjects lice free at each of the intermediate evaluations (Day 1, Day 7) | Day 1, Day 7
  Secondary outcome involved the cure rate (%) in each treatment group, following one application of the specific test product, as assessed 24h post treatment (day 1) and on day 7 (prior to the second treatment).

OTHER OUTCOMES:
Eye irritation | Day0, Day 1, Day7, Day10
  As part of the evaluation of the safety profile of both test products, eye irritation has been evaluated at day 0 (prior to and after first treatment), day 1 (24h after the first treatment), day 7 (prior to and after second treatment) and day 10, respectively.
Scalp condition | Day0, Day1, Day7, Day10
  As part of the evaluation of the safety profile of both test products, scalp condition has been evaluated at day 0 (prior to and after first treatment), day 1 (24h after the first treatment), day 7 (prior to and after second treatment) and day 10, respectively.
Adverse events collection | Day 0, Day1, Day7, Day10
  Adverse events have been collected from the initial application of test product until completion of the final follow-up visit (day 10). For any adverse event, date of onset, intensity, seriousness and causal relationship to the study treatment have been recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Serrano, Principal Investigator — Lice Source Services
Locations (1):
- Lice Source services Inc, Plantation, Florida, United States

REFERENCES:
- [Background] Barker SC, Burgess I, Meinking TL, Mumcuoglu KY. International guidelines for clinical trials with pediculicides. Int J Dermatol. 2012 Jul;51(7):853-8. doi: 10.1111/j.1365-4632.2011.05446.x. PMID 22715834